CLINICAL TRIAL: NCT03553121
Title: Jinekolojik Kanserler Nedeni Ile Opere Edilen Hastalarda Preoperatif yürümenin Postoperatif Barsak fonksiyonlarına Etkisi
Brief Title: Preoperatively Walking's Effect of Postoperative Bowel Functions in Patient With Gynecologic Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017/223
Record Dates: First submitted 2018-05-27; First posted 2018-06-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Bowel Functions
Keywords: gynecologic cancer; postoperative bowel function; walking; debulking
MeSH Terms: interventions — Walking

STUDY DESIGN:
Intervention Model Description: walking preoperatively not walking preoperatively
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Doctor who evaluate bowel function will not know whether patients walked or not
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walk preoperativelying (Active Comparator): Patients will be operated gynecologic cancers and have American Society of Anesthesia score 1 or 2. Subjects will walk during one hour with average speed 3 km/hour 12 hour before surgery.
  Interventions: Other: walking
- not walking preoperatively (Active Comparator): Patients will be operated gynecologic cancers and have American Society of Anesthesia score 1 or 2. Subjects will not walk preoperatively.
  Interventions: Other: walking

INTERVENTIONS:
Other: walking — walking and not walking

SUMMARY:
Preoperative walking's effect of postoperative bowel functions ASA 1 or 2 in patient with gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

* patients with gynecological cancer ASA score 1 or 2 via laparascopy or laparatomy

Exclusion Criteria:

* ASA score >2 orthopedic problems ileostomy or colostomy >24 hours stay in intensive care unit early postoperative complications (relaparotomy, massive blood transfusion)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
the time to the first passage of flatus after surgery | 6 hours- 5 days
  Doctor will detect the time with auscultation

SECONDARY OUTCOMES:
the time to first defecation | 6 hours- 7 day
  Doctor will detect the time with auscultation
time to first bowel movement | 6 hours- 5 days
  Doctor will detect the time with auscultation

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gungorduk K, Ozdemir IA, Gungorduk O, Gulseren V, Gokcu M, Sanci M. Effects of coffee consumption on gut recovery after surgery of gynecological cancer patients: a randomized controlled trial. Am J Obstet Gynecol. 2017 Feb;216(2):145.e1-145.e7. doi: 10.1016/j.ajog.2016.10.019. Epub 2016 Oct 22. PMID 27780709
- [Derived] Ozdemir IA, Comba C, Demirayak G, Gulseren V, Erdogan SV, Aslanova F, Afsar S, Gungorduk K. Impact of pre-operative walking on post-operative bowel function in patients with gynecologic cancer. Int J Gynecol Cancer. 2019 Oct;29(8):1311-1316. doi: 10.1136/ijgc-2019-000633. Epub 2019 Jul 19. PMID 31326951